CLINICAL TRIAL: NCT05886712
Title: Improving Equitable Access to Naloxone to Prevent Opioid Overdose Deaths Within Syringe Service Programs
Brief Title: Improving Access to Naloxone to Prevent Opioid Overdose Deaths (SAIA-Naloxone)
Acronym: SAIA-N
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: University of California, San Diego (Other); Heluna Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 00021706
Record Dates: First submitted 2023-05-12; First posted 2023-06-02 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Overdose; Implementation as Usual
MeSH Terms: conditions — Drug Overdose | interventions — Naloxone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAIA-Naloxone (Experimental): SAIA-Naloxone is an intervention that facilitates an organizational SSP level analysis of naloxone delivery by assigning a trained SAIA-Naloxone coach to apply tools and techniques and engage staff to define barriers, identify solutions, and evaluate their success in cycles until achieving desired change regarding naloxone distribution. Coaches will meet with SSPs twice per month for the first 3 months and once per month for the remaining 9 months during the 12-month intervention period.
  Interventions: Other: Naloxone
- Implementation as Usual (Other): SSPs randomized to the IAU arm will not receive support to improve naloxone distribution. SSPs in California have already adopted naloxone distribution. The investigators are therefore testing the ability of SAIA-Naloxone to optimize naloxone distribution within SSPs. Accordingly, IAU is characterized by the absence of SAIA-Naloxone with the goal of comparing whether SAIA-Naloxone improves SSPs' Naloxone distribution.
  Interventions: Other: Usual intervention

INTERVENTIONS:
Other: Naloxone — Naloxone
  Arms: SAIA-Naloxone
Other: Usual intervention — usual administered drug for overdose
  Arms: Implementation as Usual

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of a multi-faceted implementation strategy, the Systems Analysis and Improvement Approach for Naloxone (SAIA-N), in syringe service programs (SSPs). The main questions it aims to answer are:

* Does SAIA-N improve naloxone distribution (number of doses, number of people receiving naloxone) compared to implementation as usual (IAU)?
* What are the costs associated with SAIA-N and how cost-effective is the strategy?

SSPs randomized to the SAIA-N arm will participate in the strategy for a period of 12-months during which they will meet 1-2 times each month with a SAIA coach who will assist the SSP in optimizing their naloxone distribution.

Researchers will compare SAIA-N to IAU to see if naloxone distribution and costs and cost-effectiveness differ by group.

DETAILED DESCRIPTION:
The investigators plan to examine SAIA-N's impact in SSPs compared to an implementation-as-usual (IAU) condition across three aims and several related hypotheses. Data collection will take place monthly across 21 months of SSP participation. These 21 months comprise a 3-month lead-in period to establish SSP outcome data characteristics, the 12-month active period during which site randomized to SAIA-N will meet with the SAIA coach, and for an additional 6 months afterward (sustainment period) to determine whether impacts are sustained.

Aim 1. This trial's first aim is to test the effectiveness of SAIA-N on improving naloxone distribution within SSPs. The investigators hypothesize that compared with SSPs receiving IAU, SSPs receiving SAIA-N will significantly increase the number of people receiving naloxone and number of naloxone doses distributed during the 12-month active period. Further, the investigators hypothesize that SSPs receiving SAIA-N will significantly increase the number of people receiving naloxone in the 6 months after the active period (the sustainment period) compared with SSPs receiving IAU.

Aim 2. This trial's second aim will estimate the cost and cost-effectiveness of SAIA-N on improving access to naloxone at SSPs, relative to IAU. The investigators hypothesize that, relative to IAU, SAIA-N will be cost-effective at increasing the number of people receiving naloxone from SSPs.

To evaluate these aims, the investigators plan a randomized controlled interrupted time series trial with 32 SSPs in California. Sixteen SSPs will be randomly assigned to the SAIA-N arm and 16 SSPs to IAU (Figure 1). SSPs randomized to the IAU arm will not receive support to improve naloxone distribution. SSPs in California have already adopted naloxone distribution. This trial therefore tests the ability of SAIA-N to optimize naloxone distribution within SSPs. Accordingly, the IAU condition is characterized by the absence of SAIA-N with the goal of comparing whether SAIA-N improves SSPs' Naloxone distribution.

The investigators' naloxone pilot study identified implementation climate and leadership engagement as important implementation determinants that can be influenced by SAIA-N and ultimately improve naloxone distribution among SSPs. Therefore, the present study assesses change in implementation climate and leadership engagement over time. The trial will first collect SSP-specific contextual data at randomization (baseline) and 12 months after randomization from all enrolled sites. The primary contact at each SSP will be asked about basic organizational characteristics (location, number of staff, budget, etc.). Next, the primary contacts as well as other staff involved with naloxone distribution at each SSP will be asked about contextual variables such as implementation climate and leadership engagement for improving naloxone distribution.

The investigators will assess SAIA-N fidelity at the specialist level. Assessment will utilize descriptive statistics such as means/medians, standard deviations/interquartile ranges, and ranges given the small sample of specialists employed by the study (n = 2). Fidelity to SAIA-N focuses on assessing the domains of content, coverage, frequency, duration, quality, and participant responsiveness of SAIA-N. To monitor fidelity, all meetings between SAIA-N specialists and SSPs will be audio recorded, and the specialist will document each meeting with an SSP in a site-specific encounter log that includes the duration of the encounter, the roles of meeting attendees, and which of the three steps the specialist completed. Study staff will rate meeting content, quality, and participant responsiveness by reviewing 20% of recorded sessions using a fidelity checklist. To assess frequency, duration, and coverage, study staff will review and assess each encounter log.

ELIGIBILITY:
Inclusion Criteria:

* SSP is located and operates in California; SSP is authorized by CDPH; and SSP has distributed naloxone to participants in the past 30 days.

Exclusion Criteria:

* SSPs who participated in the SAIA-Naloxone pilot study (n = 2) or do not distribute naloxone (currently n = 0)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Reach (Aim 1) | 21 months
  Number of participants screened for naloxone engagement, while accounting for the total number of participants who present for services
Fidelity (Aim 1) | 21 months
  Number of people who receive naloxone, while accounting for the total number of SSP participants screened for naloxone distribution
Cost (Aim 2) (Substance Abuse Services Cost Analysis Program (SASCAP)) | 18 months
  Dollar amount of cost estimates associated with SAIA-N at the SSP level
Cost-effectiveness (Incremental Cost-effectiveness Ratio (ICER)) | 18 months
  The ratio of the difference in costs to the difference in outcomes between study groups

CONTACTS AND LOCATIONS:
Locations (1):
- RTI International, Berkeley, California, United States

IPD SHARING:
Plan to Share IPD: No